CLINICAL TRIAL: NCT02621996
Title: Hammock Positioning's Influence on the Electromyographic Activity in the Flexor Muscles in Newborn Preterm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Bruna Jardim Ferraz da Silva, Physiotherapist (master student), Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 44943415.5.0000.5208
Record Dates: First submitted 2015-11-24; First posted 2015-12-04 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Preterm Birth
Keywords: Surface Electromyography; Hypotonia; Patient Positioning
MeSH Terms: conditions — Premature Birth; Muscle Hypotonia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hammock group (Experimental): PN who will be positioned in hammock inside the incubator will be with the high trunk to about the 30th, and will be used a roll of restraint in the neck by keeping a slight lordosis to avoid suffocation risks. In two days of placement, should remain about 8 hours in the hammock, being removed during cleaning procedures, diet and medical evaluation and then immediately replaced in the hammock. The alternation of decubitus (right side, supine and left lateral) should be performed whenever the child is manipulated for these procedures.
  Interventions: Device: hammock
- control group (Active Comparator): In the control group, the position will follow the routine procedure of the Hospital Barão de Lucena, consisting of the use of restraint nests "U", made with rolled sheet placed on the mattress of the incubator and covered by another sheet. The control group incubators will also be inclined at 30 ° as routine service. During the 8 position, switching the supine will also be held, side left and side right after the baby handling to cleaning procedures, diet and medical evaluation.
  Interventions: Device: containment nest

INTERVENTIONS:
Device: hammock — PN who will be positioned in hammock inside the incubator will be with the high trunk to about the 30th, and will be used a roll of restraint in the neck by keeping a slight lordosis to avoid suffocation risks. In two days of placement, should remain about 8 hours in the hammock, being removed during cleaning procedures, diet and medical evaluation and then immediately replaced in the hammock. The alternation of decubitus (right side, supine and left lateral) should be performed whenever the child is manipulated for these procedures.
  Arms: Hammock group
Device: containment nest — In the control group, the position will follow the routine procedure of the Hospital Barão de Lucena, consisting of the use of restraint nests "U", made with rolled sheet placed on the mattress of the incubator and covered by another sheet. The control group incubators will also be inclined at 30 ° as routine service. During the 8 position, switching the supine will also be held, side left and side right after the baby handling to cleaning procedures, diet and medical evaluation.
  Arms: control group

SUMMARY:
The individual who is born premature, in addition to a CNS still in accelerated training suffers early loss of intrauterine restraint, conditions that promote hypotonia characteristic of premature birth. Given this hypotonia associated with musculoskeletal immaturity when improperly positioned in the incubator for an extended period, the PN can develop joint contractures and postural imbalances that, in most cases, are transitory, however can become persistent, causing delay in their Motor development. The aim of this study is to analyze the influence of the positioning of preterm infants in the incubator hammock on the tone and the myoelectric activity of the rectus abdominis flexor muscles, biceps and hamstrings. Study type controlled, randomized, double-blind, to be carried out from November 2015 to April 2016 will be obtained two groups, control (in containment nest "U") and experimental (with hammock) to from randomized samples with premature births in Barao de Lucena Hospital or the Hospital das Clinicas, UFPE, the Intermediate Care Units (ICU) Neonatal. The sample will consist of 30 premature. To collect, pulse oximeter will be used, electromyography, neurological testing Dubowitz and recording behavioral responses. Each baby will be accompanied for about 8 hours daytime placement for two days and three evaluations performed.

DETAILED DESCRIPTION:
The study population will consist of moderately preterm newborns, attended by SUS, admitted to the NICU of HBL or HC UFPE. From randomized samples with preterm infants born in the HBL or HC, and are admitted to the NICU, will be obtained two groups, one for positioning in hammock (experimental group) and the other in incubator containment nest "U" ( group control). The sample will consist of 30 premature babies, 15 in each group. The allocation of the PN is made in two blocks, using the site randomization.com, so that the block 1 corresponds to the group with hammock and positioning block 2, the group subjected to the usual positioning in the incubator, which at the study site it is "containment nest in U". The recruitment of premature will be conducted by researcher 1, which will identify premature the NICU potentially eligible for the study, invite the parents or guardians to sign the consent form and clear, and then make the screening (inclusion) of the truly eligible babies after filling in a checklist of eligibility criteria, always registering why exclude the other. Then, the PN will be wrapped in a sheet and carried by the investigator 1 to the support area of neonatal sector, located within the NICU, and where they will be placed on the counter, a mattress (incubator) and electromyography to carry out the assessments. Since each premature will be submitted to reviews of protocol only when alert according to the state 4 or 5 (warning with little activity and alert to activity) of the Brazelton scale, evaluations will be carried out between meals, avoiding the baby stay angry or sleepy. This procedure will be followed regardless of the position that the baby will be submitted later. In the event, the evaluation will be interrupted, and the baby will be taken back to the incubator, receiving the assistance that is required, and will be excluded from the study. The electromyographic and clinical evaluations will be conducted by researcher 1, preventing the masking at this stage. The results obtained in the evaluations (global posture, gathering maneuvers arm and popliteal angle, via video recording, and the electromyographic signal) will be analyzed by researchers 2 and 3, blind research. The EMG will be made via a portable electromyography surface mark with four channels, which will be connected to a laptop, and double electrode surface, specially developed for use in EMG, disposable, adhesive gel Ag conductor / AgCl, intended for clinical and research use. According to SENIAM recommendations (EMG Surface European consortium for the Non-Invasive Assessment of Muscles), the pads will be fixed between the motor point and the tendon of the flexor muscles: rectus abdominis, biceps and hamstrings, and the electrode reference on the left lateral malleolus. Three channels will be used to record the electrical activity unilateral (right of all PN) and simultaneously in the three above-mentioned places, so that the spontaneous muscle activity baby is captured under the same conditions. The PTN will be submitted for evaluation by surface EMG while simultaneously performed the clinical evaluation of tone with the neurological test Dubowitz. It will only be applied to size of that test by referring to the tone match the focus of this research, and only the chosen sub-items that do not require much manipulation premature. These sub-items refer to the observation of global postural baby standard (which observe the legs and the upper to the trunk in the supine position), the arms collection operation (in which it analyzes the by rapid extension muscle strength elbow, and elbow flexion speed and angle he takes after three seconds long maintained the elbow), and popliteal angle (baby knee is positioned over the abdomen and exercises to gentle pressure with the index finger behind the ankle in order to increase the popliteal angle, the maximum angle observing obtained. Test up one leg at a time). Thus, after placement of the electrodes, it will initially be observed and recorded the signal picked up by EMG of the rectus abdominis muscles, biceps and hamstrings for 30 seconds, representing the muscle tone baby home. Simultaneously to this first record in the EMG, the researcher will make the clinical evaluation of the tone by observing the posture of premature standard. Then, still using the EMG in association with the Dubowitz Test, evaluation of the maneuvers of the popliteal angle and gathering arms are made that lead to be performed 30 seconds each. Similarly, in parallel to this clinical evaluation of tone, will be made in the records EMG muscle activity of the biceps and hamstrings related to muscle resistance to stretching caused the Dubowitz test. All evaluations of muscle activity (EMG and clinical) will be recorded on video using a digital camera Sony® brand (model 1000 Cyber Shot 7.2 Mega Pixels), attached to a tripod positioned in order to capture the image of the entire PN body, so researchers can analyze 2 and 3 evaluation results, but also so that we can resolve any doubt about the future evaluations. After the evaluations, the researcher first position the PN in hammock or incubator containment nest "U", according to the randomization envelope content to it corresonding. The hammock was made of knitted fabric (100% cotton) for improved tactile comfort and prevent allergic reactions in the baby, and its dimensions follow the determinations that are in the process of patenting requested by Roberta Tenorio and Roberta Bione the National Institute of Industrial Property (INPI) in 2014, with number 19140000184 protocol and order number BR 20 2014 017 809 6. In the control group, the position will follow the routine procedure of HBL and HC, which is the use of containment nests "U" , made with rolled sheet placed on the mattress of the incubator and covered by another sheet. To identify if there was adaptation of premature positioning, physiological parameters (RR, HR and SaO2) and motor behavior (approach reactions and Withdrawal) shall be observed and recorded 5 minutes before the positioning in the hammock or incubators containment nest "U" immediately following (1 minute), after 5minutes and 10 minutes. The behavioral state of the newborn will be given by the presence or absence of specific movements welfare indicators (Approach reactions - hands to her mouth / face, holding hands, gripping motion, curling up on itself); and specific movements of stress indicators (Withdrawal reactions - aircraft wing, greeting, removal of the fingers, sitting in the air, arching). If the baby does not display any of these reactions at predefined times, the comfort will be checked only by physiological indicators. HR and SaO2 will be obtained by the pulse oximeter, and the FR will be obtained by the number of breaths per minute count made by the researcher 1. In order to detect any complications during the positioning, continuous monitoring of physiological parameters will be baby both by the researcher as one by the nursing staff of the NICU as routine neonatal sector. If there apnea situations, desaturation or no adjustment to the positioning in the hammock, the baby will be removed from this position and use the hammock will be discontinued, but should be placed in an incubator with containment nest "U" (routine neonatal HBL sector and HC), excluding the study of preterm infants and considering it as sample loss. The first stage assessment will be before the positioning, being named T0. At the end of about 8 positioning daylight hours, babies are taken from the hammock, being positioned according to routine neonatal sector (in containment nest "U" in the incubator) for the nighttime. All of the protocol tone evaluations will also be repeated the next day, 24 hours after the beginning of the positioning, both for the group that was placed in the hammock in the group that was placed in the incubator containment nest "U". This second assessment will be called T1. Again, after about 8 hours of daytime position, the baby will be removed from the hammock or position "U" for the nighttime. The final evaluation will take place the next morning, approximately 48 hours after the start of positioning hammock or containment nest, a time called T2. Also, all revaluations will be filmed for any questions that may arise.

ELIGIBILITY:
Inclusion Criteria:

* Be moderate preterm infants born with gestational ages between 31-35 weeks;
* Postnatal age from 48 hours to one week of life;
* Clinical Stability: respiratory rate between 30-60 rpm, heart rate between 120-160 bpm, oxygen saturation (SaO2) above 89%, the absence of signs of respiratory distress (Silverman-Andersen Bulletin), no cyanosis or pallor and pain / discomfort;
* Appropriate behavioral State: State 4 (inactive alert) or 5 (active alert) Brazelton

Exclusion Criteria:

* APGAR less than 7 at 5˚ minute;
* Rating as small for gestational age (SGA), according to gestational age ratio chart with birth weight;
* Being in use of drugs that interfere with the state of consciousness, as sedatives;
* preterm infants undergoing phototherapy, oxygen therapy or venous access;
* preterm infants undergoing mechanical ventilation;
* Intracranial hemorrhage grade III or IV or periventricular leukomalacia (diagnosed by ultrasound transfontanellar recorded in medical records);
* CNS infection (meningitis and encephalitis);
* seizure of History;
* Necrotizing enterocolitis at the time of examination;
* Congenital malformations, genetic syndromes, neurological disorders or diagnosed congenital STORCH infectious diseases (syphilis, toxoplasmosis, rubella, cytomegalovirus and herpes).

Ages: 48 Hours to 1 Week | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-03 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Changes on Root Means Square | 72 hours
  The evaluation with the EMG, the record average amplitude will be made of myoelectric signals in microvolts for 30 seconds, with the baby in spontaneous movement in the supine position for 30 seconds while the implementation of gathering maneuver arm, and 30 seconds while it is performed the maneuver of the popliteal angle.
  The electromyographic signals are picked up by electrodes, amplified and filtered in order to clear the most of the noise signal. For processing the data, the Miographic (Miotec Biomedical Equipment-Brazil) software, which allows the signal representation in Root Mean Square (RMS) is used.
Changes on muscle tone | 72 hours
  The clinical evaluation of tone will be realized with the neurological test Dubowitz. Initially, the researcher will make the clinical evaluation of the tone by observing the posture of premature standard. Then, the evaluation of the maneuvers of the popliteal angle and gathering arms are made that lead to be performed 30 seconds each. This clinical evaluation of tone will measure the muscle resistance to stretching and the final angles of the elbow and knee right caused the Dubowitz test.
  Clinical evaluation of the test tone with neurological Dubowitz, raw scores are generated (1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5 to 5) for each sub-item (posture global, gathering maneuver arm, right popliteal angle), which will be converted into qualitative scores (1 = "normal tone", 0.5 = "border" and 0 = "abnormal"), according to gestational age at birth , according to the conversion table raw scores of Dubowitz.

SECONDARY OUTCOMES:
Changes on behavioral state | 5 minutes before positioning and 1 minute, 5 minutes, and 10 minutes after positioning" minutes
  The behavioral state of the newborn will be given by the presence or absence of specific movements welfare indicators (Approach reactions - hands to her mouth / face, holding hands, gripping motion, curling up on itself); and specific movements of stress indicators (Withdrawal reactions - aircraft wing, greeting, removal of the fingers, sitting in the air, arching). Every move will be coded as present (1) or absent (0) during positioning with hammock. The behavioral state is observed and recorded 5 minutes before the positioning in the hammock or incubators containment nest "U" immediately following (1 minute), after 5minutes and 10 minutes.
  In cases of signs of stress prevail after placement in hammock, the RN will be removed from this position and use the hammock will be discontinued, but should be placed in an incubator with containment nest "U" (routine neonatal sector Barão de Lucena hospital), excluding the study of preterm infants.

OTHER OUTCOMES:
Changes on heart rate | 5 minutes before positioning and 1 minute, 5 minutes, and 10 minutes after positioning" minutes
  The heart rate is obtained by the pulse oximeter, being observed and recorded 5 minutes before the positioning in the hammock or incubators containment nest "U" immediately following (1 minute), after 5minutes and 10 minutes. The PN must present heart rate between 120-160 bpm in the predefined times so that there is clinically stable.
Changes on respiratory rate | 5 minutes before positioning and 1 minute, 5 minutes, and 10 minutes after positioning" minutes
  Respiratory rate is obtained by counting the number of breaths per minute taken by researcher 1, being observed and recorded 5 minutes before the positioning in the hammock or incubators containment nest "U" immediately following (1 minute), after 5minutes and 10 minutes. The PN must present respiratory rate 30-60 rpm in the predefined times so that there is clinically stable.
Changes on oxygen saturation | 5 minutes before positioning and 1 minute, 5 minutes, and 10 minutes after positioning" minutes
  Oxygen saturation is obtained by the pulse oximeter, being observed and recorded 5 minutes before the positioning in the hammock or incubators containment nest "U" immediately following (1 minute), after 5minutes and 10 minutes. The PN must present peripheral oxygen saturation (SaO2) above 89% in the predefined times so that there is clinically stable.

CONTACTS AND LOCATIONS:
Overall Officials: Karla F Lambertz, PhD, Study Director — Universidade Federal de Pernambuco; Carine Wiesiolek, PhD, Study Chair — Universidade Federal de Pernambuco
Locations (1):
- Hospital Barão de Lucena, Recife, Pernambuco, Brazil